CLINICAL TRIAL: NCT04751903
Title: The Effect of Oral Motor Stimulation on Feeding and Sucking in Preterm Infants
Brief Title: Feeding and Sucking in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Şenay ARAS DOĞAN, Assistant Professor, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 216S081; 216S081 (Other Grant/Funding Number: The Scientific and Technological Research Council of Turkey)
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Preterm Birth Complication; Breast Feeding
Keywords: Feeding; Sucking success; Oral motor stimulation; Preterm infant
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Intervention Model Description: The study was conducted as the randomized controlled and double-blind experimental trial. This study was guided by the CONSORT checklist
Who Masked: Participant
Masking Description: The study was conducted at neonatal intensive care unit (NICU) of the university hospital located in eastern Turkey between May 5th, 2017 and March 19th, 2018. The preterm infants were randomly allocated to two groups, experimental group and control group, by a computer-generated number table. The sample consisted of 77 preterm infants (39 in the experimental group and 38 in the control group) who met the inclusion criteria. The gestational weeks when babies are born were grouped as follows: 29-30 weeks, 31-32 weeks, and 33-34 weeks. In this study, only one researcher (1st author) who was not included in the intensive care team administered OMS to all the infants. Thus, the families and the NICU team were double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral motor stimulation (Experimental): After the infants were assessed by a neonatologist, Oral motor stimulation was administered to the experimental group thrice a day (at 9:00, 12:00, 15:00 hours) for 15 minutes right before feeding, over a 14-day period.
  Interventions: Behavioral: oral motor stimulation
- Control group (No Intervention): The preterm infant' the control group were only fed by the researcher thrice a day (at 9:00, 12:00, 15:00 hours) over a 14-day period.

INTERVENTIONS:
Behavioral: oral motor stimulation — Oral motor stimulation (OMS) is defined as the sensorial stimulation of cheek, lip, jaw, upper-lower gum, internal cheek, tongue and soft palate that affects the physiology of oropharyngeal mechanisms and develops feeding functions.It took 15 minutes to apply the OMS by lightly touching their cheeks, lips, gums, and tongue with fingertips for the first 12 minutes, followed by letting the infant suck on a pacifier for the remaining 3 minutes. OMS used as an alternative or supplementary early intervention strategy to develop oral feeding skills in preterm infants.
  Arms: Oral motor stimulation

SUMMARY:
This study aimed to determine the effect of oral motor stimulation (OMS) in preterm infants for successful feeding and sucking.

DETAILED DESCRIPTION:
In recent years, with advances in methods of neonatal resuscitation and caring methods, the survival rate of preterm infants has gradually increased. Sucking, swallow and respiratory dysfunction are widespread complications in the preterm infants that reason oral feeding difficulties. Safe and successful oral feeding requires proper maturation of sucking, swallowing, and respiration. The development of behaviors necessary for safe and successful nutrition begins long before birth. Jaw movements begin to be seen in the intrauterine 11th week. But sucking-swallowing-respiratory coordination is not sufficiently developed before 34 weeks of gestation. For this reason, preterm babies at the greater gestational week usually show more developed and consistent feeding skills. Maternal breast milk is best for neurodevelopment in preterm infants. Achieve oral feeding and maternal breast milk as early as possible is beneficial for preterm infants.

Oral motor stimulation (OMS) is defined as the sensorial stimulation of cheek, lip, jaw, upper-lower gum, internal cheek, tongue and soft palate that affects the physiology of oropharyngeal mechanisms and develops feeding functions. OMS used as an alternative or supplementary early intervention strategy to develop oral feeding skills in preterm infants. Previous studies have indicated that the use of OMS during or before the transition to oral feeding may not only have positive effects on the preterm infants' feeding behaviors but also enhance their general clinical course. Preterm infants who suffer from oral feeding problems often experience longterm health problems and delayed discharge from the hospital. A more effective feeding decreases adverse outcomes by decreasing hospital stays.

Preterm infants are required to prolonged NICU stay in order to stabilized, feeding, and gain optimal weight. Increasing prematurity and reduced birth weight lead to extensive resource utilization. In addition all nutritional options except breast milk increase the cost. OMS can develop sucking success and provide early oral feeding. Thus nurse labor and hospital costs may decrease and OMS can be a cost-effective application.

,

ELIGIBILITY:
Inclusion Criteria:

* Born between 29th and 34th gestational weeks, based on the mother's last menstruation date,
* Percentile measurements consistent with their gestational week measurements,
* Stable vital signs,
* APGAR scores between 4 and 10 in the 1st and 5th minutes,
* Stable for 48 hours after having received mechanical ventilation and/or continuous positive airway pressure,
* Being breastfed,
* Mother's eagerness to breastfeed the infant,
* Voluntary participation of parents in the study.

Exclusion Criteria:

* Suffered from severe asphyxia,
* Born with a low birth weight according to gestational week,
* Have intraventricular bleeding,
* With a congenital anomaly,
* Babies without their mother.

Ages: 29 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
LATCH Breastfeeding Assessment Tool | 36th gestational week , 5 minute
  It was developed by Jensen, Wallace, & Kelsay (1994). Demirhan (1997) conducted its Turkey validity test and revealed that it is a reliable and easy-to-use scale. Each criterion is rated in the point range of 0-2 points. Breastfeeding is then assessed based on the sum of these scores. The highest and lowest scores of the tool are 10 and 0, respectively, and higher scores signify breastfeeding/sucking success.
body weight | 36th gestational week ,3 minute
  The baby's body weight is weighed in grams with a digital scale.
length | 36th gestational week,1 minute
  The baby's length is measured in cm with a tape measure.
head circumference | 36th gestational week ,1 minute
  The baby's head circumference is measured in cm with a tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: Ayda ÇELEBİOĞLU, Prof., Principal Investigator — Mersin Univers; Kadir Şerafettin TEKGÜNDÜZ, Assoc. Prof, Principal Investigator — Ataturk University
Locations (1):
- Bozoku, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Aguilar-Rodriguez M, Leon-Castro JC, Alvarez-Cerezo M, Aledon-Andujar N, Escrig-Fernandez R, Rodriguez de Dios-Benlloch JL, Hervas-Marin D, Vento-Torres M. The Effectiveness of an Oral Sensorimotor Stimulation Protocol for the Early Achievement of Exclusive Oral Feeding in Premature Infants. A Randomized, Controlled Trial. Phys Occup Ther Pediatr. 2020;40(4):371-383. doi: 10.1080/01942638.2019.1698688. Epub 2019 Dec 9. PMID 31814522
- [Background] Bache M, Pizon E, Jacobs J, Vaillant M, Lecomte A. Effects of pre-feeding oral stimulation on oral feeding in preterm infants: a randomized clinical trial. Early Hum Dev. 2014 Mar;90(3):125-9. doi: 10.1016/j.earlhumdev.2013.12.011. Epub 2014 Jan 23. PMID 24461572
- [Background] Coker-Bolt P, Jarrard C, Woodard F, Merrill P. The effects of oral motor stimulation on feeding behaviors of infants born with univentricle anatomy. J Pediatr Nurs. 2013 Jan;28(1):64-71. doi: 10.1016/j.pedn.2012.03.024. Epub 2012 Apr 10. PMID 22497742
- [Background] Ghomi H, Yadegari F, Soleimani F, Knoll BL, Noroozi M, Mazouri A. The effects of premature infant oral motor intervention (PIOMI) on oral feeding of preterm infants: A randomized clinical trial. Int J Pediatr Otorhinolaryngol. 2019 May;120:202-209. doi: 10.1016/j.ijporl.2019.02.005. Epub 2019 Feb 5. PMID 30851536